CLINICAL TRIAL: NCT04873206
Title: Diagnostic and Prognostic Value of PTEN Expression in Functional and Pathological Endometrial Biopsies.
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Maisa Hashem Mohammed, lecturer of pathology, Sohag University
Other Study IDs: Soh-Med-21-04-29
Record Dates: First submitted 2021-04-30; First posted 2021-05-05 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Endometrial Hyperplasia; Endometrial Adenocarcinoma
Keywords: PTEN.; Endometrial Hyperplasia.; Endometrial Carcinoma
MeSH Terms: conditions — Endometrial Hyperplasia; Endometrial Neoplasms | interventions — Immunohistochemistry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — specimens fixed in Formalin and embedded in Parraffin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Functional/ Cyclical Endometrial group.: cases of normal endometrium will be obtained from hystrectomy specimens done for causes other than hyperplasia or adenocarcinoma, for example; uterine fibroids, uterine prolapse.
  Interventions: Other: routine stain by H&E.
- Hyperplastic Endometrial group.: cases of endometrial hyperplasia obtained by D&C or hystrectomy will be stained by H&E stain and categorized into typical or atypical hyperplasia.
  Interventions: Other: routine stain by H&E.
- Primary Endometrial Adenocarcinoma group.: cases of primary endometrial adenocarcinoma obtained by D&C or hystrectomy operations
  Interventions: Other: routine stain by H&E.

INTERVENTIONS:
Other: routine stain by H&E. — formalin fixed, Parraffin embedded endometrial tissues will be sectioned and get stained by the routine Haematoxalin and Eosin stain in addition to immunohistochemical staining by anti-human PTEN antibody.
  Other Names: Immunohistochemistry.

SUMMARY:
endometrial hyperplasia may progress to endometrial adenocarcinoma. the exact possibility of such progression is not determined. there a need to detect biological markers that can help in detecting high risk cases of patients with endometrial hyperplasia that may progress to endometrial adenocarcinoma. PTEN is a tumor suppressor gene that inhibit cell migration, proliferation and may induce apoptosis in damaged cells. variable expression of PTEN in functional, hyperplastic and neoplastic endometrial tissues may be of great help in detecting cases of hyperplasia that may progress to endometrial adenocarcinoma.

DETAILED DESCRIPTION:
Adenocarcinoma of the endometrium is the most prevalent invasive tumor of female genital tract. Endometrial carcinoma is divided to 2 different types as regards to genitical and phenotypical features, type I endometrial carcinoma represents more than three quarters of all cases. Type I is inevitably preceded by hyperplastic changes in the endometrium. However, the malignant potential of endometrial hyperplasia to carcinoma is markedly variable and subjected to interobserver variations. Determine of novel biological markers for detection of precancerous endometrial hyperplasia that may proceed to endometrial adenocarcinoma is a must. PTEN is a tumor suppressor gene. it inhibits cell mitosis and migration. PTEN induce the damaged cells to pass in apoptosis. Low levels of PTEN expression noted in many human malignancies as melanoma, mammary and ovarian carcinomas.

The aim of this study is to evaluate the expression of PTEN (by immunohistochemistry) in different endometrial biological conditions as endometrial hyperplasia and primary endometrial adenocarcinoma specimens, and correlate that expression to PTEN expression in physiological endometrial specimens.

ELIGIBILITY:
Inclusion Criteria:

* all cases of endometrial biopsies and hystrectomy specimens diagnosed as endometrial hyperplasia and/or primary endometrial adenocarcinoma.
* all cases of normal endometrium obtained from hystrectomy specimens due to other pathological conditions as prolapsed uteri, uterine leiomyoma and adenomyosis.

Exclusion Criteria:

* autolysed samples, very tiny specimens cervical tissues and specimens with histological picture of endometritis.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: endometrial specimens and hystrectomy operations will be done in Gyn&Obs Department of Sohag University Hospital and will be prepared in formalin-fixed, Parraffin-embedded blocks. endometrial blocks will be sectioned and stained by H&E stain. from the same blocks, corresponding tissue sections will be staine immunohistochemically by anti-human PTEN antibodies.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Investigating the Immunohistochemical Expression of PTEN in Different Endometrial Biopsies. | June, 2021
  cases of primary endometrial carcinoma and complex endometrial hyperplasia should express mutant form of PTEN compared to functional and simple hyperplastic endometrial tissues.

CONTACTS AND LOCATIONS:
Overall Officials: Maisa H Mohammed, MD, Principal Investigator — a lecturer of pathology, Sohag faculty of medicine
Locations (1):
- Maisa Hashem Mohammed, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided